CLINICAL TRIAL: NCT07400120
Title: Enhanced Post-Licensure Safety Surveillance Study of the Recombinant Acellular Pertussis Vaccine (aP), VacPertagen, in Thailand
Brief Title: Safety Monitoring of VacPertagen Vaccine in Thailand
Acronym: PERTg001
Status: Completed | Type: Observational
Sponsor: BioNet-Asia Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PERTg001
Record Dates: First submitted 2026-01-14; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pertussis (Whooping Cough)
Keywords: Pertussis
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VacPertagen recipients: Vaccinees consist of adults including the elderly and pregnant women in private and government hospitals and clinics located in the central, eastern, northern, and southern regions of Thailand.

SUMMARY:
In compliance with Thailand's conditional approval requirements, this prospective, observational study is designed to actively monitor the safety of VacPertagen vaccine. Healthcare professionals (HCPs) prescribing or administering the vaccine are recruited from hospitals and clinics across central, eastern, southern and northern Thailand. Adverse events following immunization (AEFIs) are reported through standardized questionnaires and modified WHO AEFI forms, enabling systematic evaluation of the vaccine's safety profile in a broader and more heterogeneous population than that assessed in pre-licensure trials.

Primary objective: To describe the post-licensure safety profile of VacPertagen in Thailand.

Secondary objective: To identify any unexpected safety signals following vaccination with VacPertagen.

DETAILED DESCRIPTION:
HCPs eligible to participate were those who prescribed or administered VacPertagen as a booster immunization in line with national guidelines. Recruitment was carried out in hospitals and clinics located in central, eastern, southern and northern Thailand. HCPs who agreed to participate were interviewed periodically regarding adverse events following immunization (AEFIs) with VacPertagen.

Data collection was performed using a standardized questionnaire administered monthly, either in person or by telephone. The questionnaire captured the number and type of AEFIs observed, along with other safety-related information.

HCPs used a modified WHO AEFI report form to document adverse events. In addition, a pregnancy safety outcome report form was developed to collect data on pregnancy outcomes among vaccinated pregnant women and their newborn. This structured approach enabled systematic monitoring of VacPertagen's safety profile in real-world conditions and ensured early identification of any unexpected safety signals.

Statistical Analysis. No formal prespecified study hypothesis was formulated. Descriptive statistics were used to summarize demographic characteristics of VacPertagen recipients, percentage of AEFIs and outcomes of pregnant women vaccinated with VacPertagen including pregnancy complications and newborn health outcomes. Overall data were analyzed using measures such as mean ± standard deviation for continuous variables and numbers with percentages for categorical variables. 95% confidence intervals were calculated for all indicators. Statistical analyses were performed using SPSS version 18 (SPSS Inc., Chicago IL).

ELIGIBILITY:
Inclusion Criteria: An HCP will be eligible for inclusion if ALL of the following criteria are met at the time of screening:

1. Has prescribed and/or administered VacPertagen to adults and adolescents in accordance with current national immunization guidelines.
2. Employed full-or part-time (> 8 hours/week) in a government or private hospital or medical clinic.
3. Available for follow-up by telephone call, email or site visit if there are missing information in the study questionnaire, to confirm the occurrence or clarify the nature of an adverse event following immunization with VacPertagen.
4. Willing and able to comply with the study procedures.

Exclusion Criteria:

* Unwilling to take part in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of a cohort of HCPs working in private and government hospitals and clinics in central, eastern, northern and southern Thailand where VacPertagen vaccine is marketed. An HCP is defined as medically qualified person, such as physician, nurse or pharmacist.
Sampling Method: Non-Probability Sample
Enrollment: 5414 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Incidence and percentage of AEFIs following vaccination with VacPertagen. | From the date of vaccination up to 30 days post-vaccination.
  Measure the frequency, categorize the types, assess the severity, and determine the causal relationship to vaccination for all AEFIs.
Incidence and percentage of pregnant women vaccinated with VacPertagen who had experienced complications during pregnancy | From administration of VacPertagen during pregnancy until delivery
  Incidence rate is defined as the number of maternal complications in 1000 vaccinees. Pregnancy complications include but are not limited to the following: pregnancy loss or stillbirth, preterm delivery (< 37 weeks of gestation), premature rupture of membranes, pregnancy-induced hypertension, pre-eclampsia/eclampsia, intrauterine growth restriction (IUGR), obstetric hemorrhage, and gestational diabetes.
Incidence and percentage of healthy and not healthy infants born to mothers who received VacPertagen during pregnancy. | From maternal vaccination during pregnancy until birth of the infant.
  Incidence rate is defined as the number of healthy and not healthy infants in 1000 infants born to mothers who received VacPertagen during pregnancy.
  This outcome assesses the health status of infants born to mothers who received VacPertagen during pregnancy. Infants will be classified at birth as healthy or not healthy based on clinical assessment and review of delivery and neonatal records.
  A healthy infant is defined as a live-born infant without any congenital anomalies, neonatal complications, or conditions requiring significant medical intervention at birth. A not healthy infant is defined as a live-born infant with at least one reported adverse neonatal outcome, including but not limited to congenital anomalies, preterm birth, low birth weight, neonatal intensive care unit (NICU) admission, or other clinically significant medical conditions identified at or shortly after birth.

SECONDARY OUTCOMES:
Incidence and percentage of unexpected serious adverse events (SAEs) following VacPertagen vaccination | From the date of vaccination up to 30 days post-vaccination for adults and up to delivery for pregnant women.
  Number and percentage of participants in each population group (adolescents, adults, and pregnant women) experiencing unexpected SAEs after VacPertagen vaccination. Events will be identified through electronic health records and classified per CIOMS/WHO definitions of SAEs and safety signals, which include any serious medical occurrence that may indicate a new potential association requiring further evaluation.
Incidence and percentage of rare adverse events following VacPertagen vaccination | From the date of vaccination up to 30 days post-vaccination for adults and up to delivery for pregnant women.
  Number and percentage of participants with medically confirmed, rare adverse events (events too uncommon to be detected in pre-licensure trials). Rare adverse event is defined as event occurring with a frequency of ≥ 1/10,000 and < 1/1,000).
Incidence and percentage of new patterns of known adverse events | From the date of vaccination up to 30 days post-vaccination for adults and up to delivery for pregnant women.
  Number and percentage of participants presenting new patterns of adverse events already associated with pertussis-containing vaccines (e.g., shifts in severity, timing, clustering). Safety signals include new aspects of known associations, per CIOMS/WHO definitions. Data will be analyzed using temporal clustering and disproportionality analysis to identify unexpected patterns following VacPertagen vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, PhD., Study Director — BioNet-Asia Co., Ltd.
Locations (1):
- BioNet-Asia Co.,Ltd., Bangkok, Bangkok, Thailand